CLINICAL TRIAL: NCT01514786
Title: Decision Aid to Technologically Enhance Shared Decision Making
Acronym: DATES
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Masahito Jimbo, MD, Clinical Associate Professor, Family Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00044733
Record Dates: First submitted 2012-01-17; First posted 2012-01-23 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Colorectal Cancer
Keywords: Colorectal Cancer; Screening; Prevention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Same information is presented in the control website as is found in the intervention website, but no interactive component: preferences and risk assessment.
- Intervention with Colorectal Website (Active Comparator): Intervention website includes an interactive component including preferences and risk assessment.
  Interventions: Behavioral: Colorectal Web

INTERVENTIONS:
Behavioral: Colorectal Web — The intervention arm will allow participants on Colorectal Web to manipulate their preferences for CRCS
  Arms: Intervention with Colorectal Website

SUMMARY:
Physicians face a challenge in promoting colorectal cancer screening (CRCS) in the face of multiple competing demands. A decision aid (DA) that clarifies patient preferences and improves decision quality could aid shared decision making (SDM) and be effective at increasing CRCS rates. However, exactly how such DA improves SDM is not clear. This 4-year R01 study funded by the National Cancer Institute seeks to provide detailed understanding of how an interactive DA affects patient-physician communication and SDM, and ultimately CRCS adherence.

DETAILED DESCRIPTION:
This two-armed randomized controlled trial (300 patients/arm) will compare Colorectal Web (CW), the interactive DA, to a non-interactive control website in ten practices in Metro Detroit. Patients will be adults aged 50 years and over, not current on CRCS. In the clinic before the patient-physician encounter, participants will complete a Patient Baseline Survey. They will be randomized to CW or the control website. Data will be collected after the patient reviews the respective website (Post-Intervention Survey), during the patient-physician encounter (digital audio recording), and after it (Post-Encounter Survey). Chart audit will be performed six months after the encounter to determine whether the patient underwent CRCS.

ELIGIBILITY:
Inclusion Criteria:

* 50-75 years of age
* not current with colorectal cancer screening
* scheduled for HME, Health Maintenance Exam, or chronic care visit with participating physician
* able to read English
* current contact information

Exclusion Criteria:

* history of colon cancer or adenomatous polyps
* history of dementia or psychosis
* contraindication to CRCS

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 570 (Actual)
Dates: Start 2012-05; Primary Completion 2014-09 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Masahito Jimbo, MD, PhD, MPH, Principal Investigator — University of Michigan
Locations (14):
- United States (14):
  - Children's and Family Medical Clinic, Allen Park, Michigan
  - Downriver Internists, Allen Park, Michigan
  - University of Michigan Family Medicine at Domino's, Ann Arbor, Michigan
  - University of Michigan Briarwood Family Medicine, Ann Arbor, Michigan
  - Dua Family Practice, Canton, Michigan
  - George C. Hawrot, MD, Dearborn, Michigan
  - Andrew Thomas, MD, Detroit, Michigan
  - Morang Chester Clinic, Detroit, Michigan
  - Rice Lanzilote & Egan, Detroit, Michigan
  - David Williams, MD, Detroit, Michigan
  - IPC - Livonia Internal Medicine, Livonia, Michigan
  - Lonnie Joe Jr. MD, Southfield, Michigan
  - Mark W. Sawka, MD, Woodhaven, Michigan
  - University of Michigan Family Medicine at Corner Health Center, Ypsilanti, Michigan

IPD SHARING:
Plan to Share IPD: Yes
Data is still being analyzed and papers written

REFERENCES:
- [Derived] Jimbo M, Sen A, Plegue MA, Hawley S, Kelly-Blake K, Rapai M, Zhang M, Zhang Y, Xie X, Ruffin MT 4th. Interactivity in a Decision Aid: Findings From a Decision Aid to Technologically Enhance Shared Decision Making RCT. Am J Prev Med. 2019 Jul;57(1):77-86. doi: 10.1016/j.amepre.2019.03.004. Epub 2019 May 23. PMID 31128959
- [Derived] Jimbo M, Kelly-Blake K, Sen A, Hawley ST, Ruffin MT 4th. Decision Aid to Technologically Enhance Shared decision making (DATES): study protocol for a randomized controlled trial. Trials. 2013 Nov 11;14:381. doi: 10.1186/1745-6215-14-381. PMID 24216139

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention With Colorectal Website
Started | 286 | 284
Completed | 286 | 284
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention With Colorectal Website | Total
Number analyzed (Participants) | 286 | 284 | 570
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 231 | 240 | 471
  >=65 years | 55 | 44 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (6.9) | 57.1 (6.8) | 57.7 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 177 | 143 | 320
  Male | 109 | 141 | 250
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 286 | 284 | 570
Participants screened for colon cancer [Count of Participants; unit: Participants] | 111 | 99 | 210

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Preferred Screening Type as Reported by Chart Audits
Description: Chart audits were conducted 6 months after the participant's study visit to determine if screening had occurred and if the type of screen was the same as the participant's preferred type of screening.
Time Frame: 6 months following intervention a chart audit will be conducted to determine if CRCS was completed.
Measure: Number; unit: participants
Arm/Group | Control | Intervention With Colorectal Website
Number analyzed (Participants) | 286 | 284
participants | 111 | 99

ADVERSE EVENTS:
Time Frame: During 2 year data collection period
Description: No difference
  This study involved participants looking at a website and completing questionnaires regarding colon cancer risks and screening. The risks of participating in these activities are no greater than participating in everyday activities. The participant who died after consenting died during knee surgery, totally unrelated to participating in the study. This was the only AE that study staff became aware of during the study period.
Arm/Group | Control | Intervention With Colorectal Website
All-Cause Mortality (participants affected / at risk) | 0/286 | 1/284
Serious Adverse Events (participants affected / at risk) | 0/286 | 1/284
Other Adverse Events (participants affected / at risk) | 0/286 | 0/284
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=286) | Intervention With Colorectal Website (N=284)
Death (General disorders) | 0 (0) | 1 (1) — Participant's death occurred during surgery totally unrelated to participation in the study. Clinic site staff member just happened to mention to research study staff this happened.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No